CLINICAL TRIAL: NCT06834490
Title: International Multicentre Randomized, Double-blind, Placebo-controlled Adaptive Design Clinical Trial to Evaluate the Safety and Efficacy of Sequential Therapy With Mexidol® Solution for Intravenous and Intramuscular Administration, 50 mg/ml (RPC PHARMASOFT LLC, Russia) and Mexidol® FORTE 250 Film-coated Tablets, 250 mg (RPC PHARMASOFT LLC, Russia) in Patients With Chronic Cerebral Ischemia (MEMO)
Brief Title: Safety and Efficacy of Sequential Therapy With Mexidol® in Patients With Chronic Cerebral Ischemia
Acronym: MEMO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pharmasoft (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MexidolMEMO2020; PHS-CICADIS-005-MEX-SOL-TAB (Other: Pharmasoft)
Record Dates: First submitted 2025-02-11; First posted 2025-02-19 (Actual); Results first posted 2025-10-06 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Chronic Cerebral Ischemia
Keywords: Chronic Cerebral Ischemia; CCI; Ischemia; Cerebral; Brain; Stroke; Cognitive; Neurobehavioral Manifestations; Neuroprotection; Mexidol; Ethylmethylhydroxypyridine Succinate; Cerebrovascular Disorders; Antioxidant Therapy; Stroke Recovery; Central Nervous System Disorders; Chronic Brain Hypoxia; Post-stroke Cognitive Impairment; Cognitive Impairment; Neurodegenerative; Neurodegenerative Processes; Neurological Rehabilitation; Oxidative Stress; Oxidative Stress Reduction; Energy Metabolism Enhancement; Central Nervous System; Cerebral Hypoxia
MeSH Terms: conditions — Ischemia; Stroke; Neurobehavioral Manifestations; Cerebrovascular Disorders; Central Nervous System Diseases; Cognitive Dysfunction; Hypoxia, Brain | interventions — emoxypine succinate; ethylmethylhydroxypyridine succinate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Main (Mexidol) (Active Comparator): Participants received Mexidol IV 500 mg (10 ml) once daily for 14 days, then Mexidol FORTE 250 orally 250 mg 1 tablet 3 times a day for 60 days
  Interventions: Drug: Mexidol
- Control (Placebo) (Placebo Comparator): Participants received Mexidol Placebo matching Mexidol IV 500 mg (10 ml) once daily for 14 days, then Mexidol Placebo matching Mexidol FORTE 250 orally 250 mg 1 tablet 3 times a day for 60 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Mexidol — 50 mg/ml IV solution, 250 mg tablets
  Other Names: Ethylmethylhydroxypyridine Succinate
  Arms: Main (Mexidol)
Drug: Placebo — Placebo IV solution, Placebo tablets
  Arms: Control (Placebo)

SUMMARY:
The purpose of this study is to evaluate safety and efficacy of sequential treatment with Mexidol® in patients with chronic cerebral ischemia (CCI).

DETAILED DESCRIPTION:
Chronic cerebral ischemia (CCI) is a cerebral vascular pathology caused by slow progressive diffuse disruption of blood flow to the brain with gradually increasing defects in its functioning. The activation of lipid peroxidation with the release of large amounts of active oxygen radicals plays the key role in the pathogenesis of ischemic disorders, which leads to the development of oxidative stress. However, traditional drug therapy, which is aimed at improving blood flow to the brain, is mainly based on drugs with psychostimulant component, and does not always prevent the increase of oxidative damage to the patients' body. That is why it is necessary to search for drugs that would correct these processes selectively. Mexidol contains ethylmethylhydroxypyridine succinate as an active substance and may be the drug of choice for the treatment of CCI patients.

ELIGIBILITY:
Inclusion criteria:

1. Patients of either sex aged from 40 to 90 years inclusive
2. MoCA scale score of 25 and lower
3. Patients meeting the criteria for the diagnosis: Mild (moderate) cognitive impairment when assessed by DSM-5.
4. Chronic Cerebral Ischemia (ICD-10 code 167.8)
5. Foci of leukoaraiosis or "silent" brain infarction documented by MRI/CT performed within the past 12 months.
6. Patients who signed an informed consent to the study participation
7. History of progressive multifocal or diffuse brain disease from 1 to 5 years
8. Patients receiving background therapy with a fixed dose and combination of drugs during the previous month, including (if indicated): antiplatelet therapy, therapy of cerebral atherosclerosis and arterial hypertension, ischemic heart disease or other chronic diseases.
9. Negative pregnancy test
10. Patients who have agreed to use a reliable method of contraception during the study participation until completion (for women of childbearing potential, including partners of study participants).
11. Patients who are able to understand all study requirements and who have consented to all the limitations imposed by the study

Exclusion Criteria:

1. Inclusion by mistake (overlooked inclusion or non-inclusion criteria)
2. Investigator's or Sponsor's decision to exclude a participant from the study due to a clinically significant protocol deviation/violation.
3. Serious adverse events or adverse events that do not meet the criteria for seriousness but may, in the investigator's opinion, be detrimental to the health or well-being of a participant if they continue participation in the study.
4. Any adverse event (which may be unrelated to the investigational drug) requiring observations, procedures, and/or medications not approved by the clinical trial protocol.
5. Participant's refusal to continue participation in the study or their lack of discipline
6. Allergic reaction to the investigational drug that requires cancelling the treatment
7. Participant's desire to terminate their participation early for any reason.
8. Loss of contact with the patient followed by failure to attend the visit.
9. The need to take therapies prohibited by this protocol: nootropic drugs, ethylmethylhydroxypyridine succinate, trimetazidine or meldonium, drugs affecting the function of the autonomic nervous system and other drugs that may, in the investigator's opinion, distort the study results.
10. Pregnancy.

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 318 (Actual)
Dates: Start 2019-11-05 (Actual); Primary Completion 2020-12-08 (Actual); Study Completion 2020-12-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alina S. Agafina, MD, Cand.Med.Sci, Principal Investigator — Saint Petersburg State Budget Healthcare Institution "City Hospital No.40 of the Kurortny District"; Elena V. Vostrikova, MD, Cand.Med.Sci, Principal Investigator — State Budget Healthcare Institution of the Nivisibirsk Region "City Hospital No.34"; Andrey M. Alasheev, MD, Dr.Med.Sci, Principal Investigator — State Budget Healthcare Institution of the Sverdlovsk Region "Sverdlovsk Regional Clinical Hospital No.1"; Marine M. Tanashyan, Prof., Dr.Med.Sci, Principal Investigator — Federal State Budget Research Institution "Research Center of Neurology"; Min G. Omelyanenko, MD, Dr.Med.Sci, Principal Investigator — Regional Budget Healthcare Institution "Ivanovo Regional Clinical Hospital"; Stanislav O. Pozdnyakov, MD, Cand.Med.Sci, Principal Investigator — OOO "Centre for Evidence-Based Medicine"; Aleksandr Y. Malygin, MD, Dr.Med.Sci, Principal Investigator — State Budget Healthcare Institution of the Yaroslavl Region "Clinical Hospital No.2"; Aida A. Yakupova, MD, Cand.Med.Sci, Principal Investigator — Federal State Budget Educational Institution of Higher Education "Kazan State Meical University"; Igor V. Litvinenko, Prof., Dr.Med.Sci, Principal Investigator — Federal State Budget Military Educational Institution of Higher Education "Military Medical Academy n.a. S.M.Kirov"; Irina G. Lukashevich, MD, Principal Investigator — Municipal Autonomous Healthcare Insitution of the Order of the Red Banner of Labour "City Clinical Hospital No.1"; Olga A. Sinitsyna, MD, Cand.Med.Sci, Principal Investigator — State Budget Healthcare Institution of the Yaroslavl Region "Clinical Hospital No.2"; Larisa A. Shchepankevich, MD, Dr.Med.Sci, Principal Investigator — Federal State Budget Research Institution "Federal Research Center for Fundamental and Translational Medicine"; Galina A. Batishcheva, Prof., Dr.Med.Sci, Principal Investigator — Private Healthcare Institution "Clinical Hospital "RR-Medicine" of Voronezh; Olga D. Ostroumova, Prof., Dr.Med.Sci, Principal Investigator — Federal State Budget Educational Institution of Further Professional Education "Russian Medical Academy of Continuous Professional Education"; Yokutkhon N. Madzhidova, Prof., Dr.Med.Sci, Principal Investigator — Centre for Neurology and Neurorehabilitation n.a. N.M.Madzhido, OOO "Neyromed Servis"
Locations (14):
- Russia (13):
  - Municipal Autonomous Healthcare Insitution of the Order of the Red Banner of Labour "City Clinical Hospital No.1", Chelyabinsk
  - Regional Budget Healthcare Institution "Ivanovo Regional Clinical Hospital", Ivanovo
  - Federal State Budget Educational Institution of Higher Education "Kazan State Medical University", Kazan'
  - Federal State Budget Research Institution "Research Center of Neurology", Moscow
  - Federal State Budget Educational Institution of Further Professional Education "Russian Medical Academy of Continuous Professional Education", Moscow
  - State Budget Healthcare Institution of the Novosibirsk Region "City Hospital № 34", Novosibirsk
  - Federal State Budget Research Institution "Federal Research Center for Fundamental and Translational Medicine", Novosibirsk
  - Federal State Budget Military Educational Institution of Higher Education "Military Medical Academy n.a. S.M.Kirov", Saint Petersburg
  - City Hospital No.40 of the Kurortny District, Sestroretsk
  - Private Healthcare Institution "Clinical Hospital "RR-Medicine" of Voronezh, Voronezh
  - OOO "Centre for Evidence-Based Medicine", Yaroslavl
  - State Budget Healthcare Institution of the Yaroslavl Region "Clinical Hospital No.2", Yaroslavl
  - State Budget Healthcare Institution of the Sverdlovsk Region "Sverdlovsk Regional Clinical Hospital No.1", Yekaterinburg
- Centre for Neurology and Neurorehabilitation n.a. N. M. Madzhido, OOO "Neyromed Servis", Tashkent, Uzbekistan

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited based on protocol requirements at 15 clinical sites between November 2019 and December 2020. The first participant was enrolled on 05 November, 2019 and the last participant was enrolled on 14 September, 2020.
Pre-assignment Details: Of 330 screened participants, 318 met inclusion criteria and were randomized to treatment.
Period: Overall Study
Arm/Group | Main (Mexidol) | Control (Placebo)
Started | 159 | 159
Completed | 157 | 155
Not Completed | 2 | 4

BASELINE CHARACTERISTICS:
Population: ITT-population was used for description of baseline measures.
Groups:
- Total: Total of all reporting groups
Arm/Group | Main (Mexidol) | Control (Placebo) | Total
Number analyzed (Participants) | 159 | 159 | 318
Age, Categorical [Count of Participants; unit: Participants] — Patients aged from 40 to 90 years inclusive were enrolled
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 104 | 99 | 203
    >=65 years | 55 | 60 | 115
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.08 (9.86) | 60.73 (9.03) | 60.44 (9.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 119 | 121 | 240
  Male | 40 | 38 | 78
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 10 | 8 | 18
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 149 | 151 | 300
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants] — Population: There were 302 participants from Russia and 16 participants from Uzbekistan. 302 plus 16 equals 318 (ITT-population).
  Participants
    Russia: number analyzed (Participants) | 151 | 151 | 302
    Russia | 151 | 151 | 302
    Uzbekistan: number analyzed (Participants) | 8 | 8 | 16
    Uzbekistan | 8 | 8 | 16
The Montreal Cognitive Assessment scores at Visit 0 (7 days before treatment) [Mean (Standard Deviation); unit: score on a scale] — The Montreal Cognitive Assessment (MoCA) is used to measure the changes in the severity of cognitive impairment at Visits 2 and 4 in comparison to Visit 0. MoCA scores range between 0 and 30. A score of 26 or over is considered to be normal. Population: The results obtained at Visit 0 were used as the reference for the estimation of the efficacy. The statistical analysis was performed for ITT-population excluding participant No. 098 whose data after the randomization visit are missing.
  score on a scale
    number analyzed (Participants) | 159 | 158 | 317
    (all) | 21.53 (2.27) | 21.80 (1.96) | 21.67 (2.13)
The SF-36 questionnaire scores at Visit 1 (Day 1 of treatment) [Mean (Standard Deviation); unit: score on a scale] — The SF-36 questionnaire has two summary measures: physical and mental health. The scoring ranges from 0 to 100. Higher scores indicate better health status. Population: The results obtained at Visit 1 were used as the reference for the estimation of the efficacy. The statistical analysis was performed for ITT-population excluding participant No. 098 whose data after the randomization visit are missing.
  score on a scale
    The SF-36 questionnaire: physical health: number analyzed (Participants) | 159 | 158 | 317
    The SF-36 questionnaire: physical health | 44.21 (8.58) | 44.12 (7.92) | 44.21 (8.28)
    The SF-36 questionnaire: mental health: number analyzed (Participants) | 159 | 158 | 317
    The SF-36 questionnaire: mental health | 44.12 (9.18) | 44.95 (9.20) | 44.51 (9.18)
The Multidimensional Fatigue Inventory scores at Visit 1 (Day 1 of treatment) [Mean (Standard Deviation); unit: score on a scale] — MFI-20 is a 20-item self-administered questionnaire designed to measure fatigue in five four-item subscales: General fatigue, Physical fatigue, Reduced activity, Reduced motivation and Mental fatigue. Population: The results obtained at Visit 1 were used as the reference for the estimation of the efficacy. The statistical analysis was performed for ITT-population excluding participant No. 098 whose data after the randomization visit are missing.
  score on a scale
    number analyzed (Participants) | 159 | 158 | 317
    (all) | 59.77 (13.35) | 58.79 (13.78) | 59.25 (13.55)
The Beck Anxiety Inventory scores at Visit 1 (Day 1 of treatment) [Mean (Standard Deviation); unit: score on a scale] — The Beck Anxiety Inventory (BAI) consists of 21 self-reported items (four-point scale) used to assess the intensity of physical and cognitive anxiety symptoms during the past week. Scores may range from 0 to 63: minimal anxiety levels (0-7), mild anxiety (8-15), moderate anxiety (16-25), and severe anxiety (26-63). Population: The results obtained at Visit 1 were used as reference for the estimation of the efficacy. The statistical analysis was performed for ITT-population excluding participant No. 098 whose data after the randomization visit are missing.
  score on a scale
    number analyzed (Participants) | 159 | 158 | 317
    (all) | 11.85 (8.11) | 11.23 (8.54) | 11.51 (8.33)
A.M.Wein's questionnaire scores at Visit 1 (Day 1 of treatment) [Mean (Standard Deviation); unit: score on a scale] — The A.M.Wein's questionnaire is used between Visit 1 and Visit 2, 4, 5. It includes 11 main signs of autonomic disorders. Each autonomic symptom is assessed using scores from 3 to 7, then the scores are summed. Scores may range from 0 to 60, higher scores mean a worse outcome. The total sum of the scores in healthy individuals should be 0-14 scores, 15-29 scores are indicative of moderate vegetative dystonia syndrome, 30 and more scores are indicative of severe vegetative dystonia syndrome. Population: The results obtained at Visit 1 were used as the reference for the estimation of the efficacy. The statistical analysis was performed for ITT-population excluding participant No. 098 whose data after the randomization visit are missing.
  score on a scale
    number analyzed (Participants) | 159 | 158 | 317
    (all) | 26.59 (13.63) | 26.28 (12.70) | 26.43 (13.13)
The Digit Symbol Substitution Test scores at Visit 1 (Day 1 of treatment) [Mean (Standard Deviation); unit: score on a scale] — The DSST is used to measure attention, processing speed and executive function. It is a pencil and paper test of psychomotor performance in which the subject is given a key grid of numbers and matching symbols and a test section with numbers and empty boxes. The test consists of filling as many empty boxes as possible with a symbol matching each number. The score is the number of correct number-symbol matches achieved in 90 s. Scores range from 0 to 100, with higher scores indicating higher cognitive function. Population: The results obtained at Visit 1 were used as the reference for the estimation of the efficacy. The statistical analysis was performed for ITT-population excluding participant No. 098 whose data after the randomization visit are missing.
  score on a scale
    number analyzed (Participants) | 159 | 158 | 317
    (all) | 32.84 (10.94) | 33.87 (12.24) | 33.36 (11.63)
The Tinetti test scores at Visit 1 (Day 1 of treatment) [Mean (Standard Deviation); unit: score on a scale] — The Tinetti test is a clinical test for the assessment of balance and gait. It has a gait score and a balance score using a 3-point ordinal scale of 0, 1 and 2. Gait is scored over 12 and balance is scored over 16 totalling 28. The lower the score on the Tinetti test, the higher the risk of falling. Tinetti test score equal or less than 18 shows high risk of fall, 19-23 scores show moderate risk of fall, and score equal or higher than 24 shows low risk of fall. Thus, min value is 0, max value is 28, higher scores mean a better outcome. Population: The results obtained at Visit 1 were used as the reference for the estimation of the efficacy. The statistical analysis was performed for ITT-population excluding participant No. 098 whose data after the randomization visit are missing.
  score on a scale
    number analyzed (Participants) | 159 | 158 | 317
    (all) | 32.64 (5.30) | 33.30 (5.23) | 32.99 (5.27)

OUTCOME MEASURES:

1. Primary Outcome: Mean Score of Montreal Cognitive Assessment (MoCA) at Visit 5 in Comparison With Reference Score at Visit 0
Description: The Montreal Cognitive Assessment (MoCA) is used to measure the degree of cognitive impairment in patients with CCI. MoCA scores range between 0 and 30. A score of 26 or over is considered to be normal. Higher score than shown at Visit 0 is expected after treatment.
Time Frame: Day 75+2 (Visit 5) compared with the baseline level (Visit 0, 7 days before treatment)
Population: The efficacy analysis was performed for ITT-population excluding participant No. 098 whose data after the randomization visit are missing.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Main (Mexidol) | Control (Placebo)
Number analyzed (Participants) | 159 | 158
score on a scale
  MoCA Scores at Visit 5 | 25.72 (2.47) | 23.95 (2.58)
  Difference in comparison with Visit 0 | 4.22 (2.59) | 2.17 (2.20)

2. Secondary Outcome: Changes in the Severity of Cognitive Impairment Assessed With the Montreal Cognitive Assessment Scale Between Visit 0 and Visits 2 and 4
Description: The Montreal Cognitive Assessment (MoCA) is used to measure the changes in the severity of cognitive impairment at Visits 2 and 4 in comparison to Visit 0. MoCA scores range between 0 and 30. A score of 26 or over is considered to be normal. Higher score than shown at Visit 0 is expected.
Time Frame: Day 14 (Visit 2) and Day 44±2 (Visit 4) compared with the baseline level (Visit 0, 7 days before treatment)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Main (Mexidol) | Control (Placebo)
Number analyzed (Participants) | 159 | 158
score on a scale
  MoCA scores at Visit 2 | 23.82 (2.28) | 23.10 (2.17)
  Difference at Visit 2 in comparison to Visit 0 | 2.30 (1.96) | 1.31 (1.64)
  MoCA scores at Visit 4 | 25.06 (2.37) | 23.75 (2.34)
  Difference at Visit 4 in comparison to Visit 0 | 3.54 (2.36) | 1.98 (2.00)

3. Secondary Outcome: Changes in Patients' Quality of Life Assessed With SF-36 Questionnaire (Physical Health)
Description: The SF-36 questionnaire is used between Visit 1 and Visits 2, 4, 5. The SF-36 questionnaire consists of eight scales yielding two summary measures: physical and mental health. To score the SF-36, scales are standardized with a scoring algorithm or by the SF-36v2 scoring software to obtain a score ranging from 0 to 100. Higher scores indicate better health status, and a mean score of 50 has been articulated as a normative value for all scales.
Time Frame: Day 14 (Visit 2), Day 44±2 (Visit 4), Day 75+2 (Visit 5) compared with the baseline level (Visit 1, Day 1 of treatment)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Main (Mexidol) | Control (Placebo)
Number analyzed (Participants) | 159 | 158
score on a scale
  SF-36: physical health (Visit 2) | 44.81 (8.28) | 44.94 (7.83)
  Difference at Visit 2 in comparison with Visit 1 | 0.60 (5.29) | 0.79 (4.53)
  SF-36: physical health (Visit 4) | 46.52 (7.90) | 46.07 (7.78)
  Difference at Visit 4 in comparison with Visit 1 | 2.35 (6.07) | 2.03 (5.60)
  SF-36: physical health (Visit 5) | 47.31 (7.96) | 46.27 (7.77)
  Difference at Visit 5 in comparison with Visit 1 | 3.08 (6.70) | 2.23 (5.79)

4. Secondary Outcome: Changes in Patients' Quality of Life Assessed With SF-36 Questionnaire (Mental Health)
Description: as for outcome 3
Time Frame: Day 14 (Visit 2), Day 44±2 (Visit 4), Day 75+2 (Visit 5) compared with the baseline level (Visit 1, Day 1 of treatment)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Main (Mexidol) | Control (Placebo)
Number analyzed (Participants) | 159 | 158
score on a scale
  SF-36: mental health (Visit 2) | 46.64 (8.91) | 46.40 (9.16)
  Difference at Visit 2 in comparison with Visit 1 | 2.52 (6.75) | 1.49 (4.70)
  SF-36: mental health (Visit 4) | 48.46 (8.74) | 47.38 (9.14)
  Difference at Visit 4 in comparison with Visit 1 | 4.30 (7.85) | 2.45 (6.46)
  SF-36: mental health (Visit 5) | 50.51 (7.96) | 48.40 (8.77)
  Difference at Visit 5 in comparison with Visit 1 | 6.36 (8.14) | 3.46 (8.05)

5. Secondary Outcome: Changes in the Severity of Asthenia Assessed With the Multidimensional Fatigue Inventory (MFI-20)
Description: The Multidimensional Fatigue Inventory (MFI-20) is used between Visit 1 and Visits 2, 4, 5. MFI-20 is a 20-item self-administered questionnaire designed to measure fatigue in five four-item subscales: General fatigue, Physical fatigue, Reduced activity, Reduced motivation and Mental fatigue. MFI-20 has an even proportion of positively and negatively worded items that are rated on a 5-point Likert scale. Subscale scores (range 4-20) are calculated as the sum of item ratings and a total fatigue score (range 20-100) is calculated as the sum of subscale scores. Higher scores indicate a higher level of fatigue.
Time Frame: Day 14 (Visit 2), Day 44±2 (Visit 4), Day 75+2 (Visit 5) compared with the baseline level (Visit 1, Day 1 of treatment)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Main (Mexidol) | Control (Placebo)
Number analyzed (Participants) | 159 | 158
score on a scale
  MFI-20 scores at Visit 2 | 56.51 (13.71) | 57.14 (13.79)
  Difference at Visit 2 in comparison with Visit 1 | -3.26 (9.58) | -1.68 (7.24)
  MFI-20 scores at Visit 4 | 53.44 (14.20) | 55.23 (14.14)
  Difference at Visit 4 in comparison with Visit 1 | -6.37 (11.61) | -3.81 (10.15)
  MFI-20 scores at Visit 5 | 51.47 (13.89) | 54.24 (14.00)
  Difference at Visit 5 in comparison with Visit 1 | -8.33 (12.68) | -4.80 (11.42)

6. Secondary Outcome: Changes in the Anxiety Level According to the Beck Anxiety Inventory
Description: The Beck Anxiety Inventory (BAI) consists of 21 self-reported items (four-point scale) used to assess the intensity of physical and cognitive anxiety symptoms during the past week. Scores may range from 0 to 63: minimal anxiety levels (0-7), mild anxiety (8-15), moderate anxiety (16-25), and severe anxiety (26-63).
Time Frame: Day 14 (Visit 2), Day 44±2 (Visit 4), Day 75+2 (Visit 5) compared with the baseline level (Visit 1, Day 1 of treatment)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Main (Mexidol) | Control (Placebo)
Number analyzed (Participants) | 159 | 158
score on a scale
  BAI scores at Visit 2 | 9.97 (8.10) | 10.08 (7.23)
  Difference at Visit 2 in comparison with Visit 1 | -1.88 (5.10) | -1.11 (5.54)
  BAI scores at Visit 4 | 8.10 (7.04) | 9.14 (7.13)
  Difference at Visit 4 in comparison with Visit 1 | -3.77 (5.09) | -2.02 (5.98)
  BAI scores at Visit 5 | 7.07 (6.42) | 8.90 (7.15)
  Difference at Visit 5 in comparison with Visit 1 | -4.70 (5.49) | -2.26 (7.10)

7. Secondary Outcome: Autonomic Changes According to the A.M.Wein's Questionnaire
Description: The A.M.Wein's questionnaire is used between Visit 1 and Visit 2, 4, 5. It includes 11 main signs of autonomic disorders. Each autonomic symptom is assessed using scores from 7 to 3, then the scores are summed. Scores may range from 0 to 60, higher scores mean a worse outcome. The total sum of the scores in healthy individuals should be 0-14 scores. 15-29 scores are indicative of moderate vegetative dystonia syndrome, 30 and more scores are indicative of severe vegetative dystonia syndrome.
Time Frame: Day 14 (Visit 2), Day 44±2 (Visit 4), Day 75+2 (Visit 5) compared with the baseline level (Visit 1, Day 1 of treatment)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Main (Mexidol) | Control (Placebo)
Number analyzed (Participants) | 159 | 158
score on a scale
  Wein's questionnaire, Visit 2 | 23.58 (13.68) | 24.11 (12.61)
  Difference at Visit 2 in comparison with Visit 1 | -3.01 (7.71) | -2.18 (8.01)
  Wein's questionnaire, Visit 4 | 21.37 (13.80) | 22.89 (12.61)
  Difference at Visit 4 in comparison with Visit 1 | -5.23 (9.19) | -3.42 (10.23)
  Wein's questionnaire, Visit 5 | 19.70 (13.92) | 22.01 (13.07)
  Difference at Visit 5 in comparison with Visit 1 | -6.76 (10.94) | -4.30 (10.81)

8. Secondary Outcome: Changes in Cognitive Impairment Assessed With Digit Symbol Substitution Test
Description: The Digit Symbol Substitution Test is used between Visit 1 and Visits 2, 4, 5. The DSST is used to measure attention, processing speed and executive function.
  It is a pencil and paper test of psychomotor performance in which the subject is given a key grid of numbers and matching symbols and a test section with numbers and empty boxes. The test consists of filling as many empty boxes as possible with a symbol matching each number. The score is the number of correct number-symbol matches achieved in 90 s. Scores range from 0 to 100, with higher scores indicating higher cognitive function.
Time Frame: Day 14 (Visit 2), Day 44±2 (Visit 4), Day 75+2 (Visit 5) compared with the baseline level (Visit 1, Day 1 of treatment)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Main (Mexidol) | Control (Placebo)
Number analyzed (Participants) | 159 | 158
score on a scale
  DSST, Visit 2 | 36.94 (10.82) | 36.33 (11.84)
  Difference at Visit 2 in comparison with Visit 1 | 4.11 (6.63) | 2.61 (7.18)
  DSST, Visit 4 | 39.80 (10.78) | 37.89 (11.78)
  Difference at Visit 4 in comparison with Visit 1 | 6.91 (8.10) | 4.24 (8.77)
  DSST, Visit 5 | 42.72 (12.53) | 39.05 (12.36)
  Difference at Visit 5 in comparison with Visit 1 | 9.84 (10.50) | 5.40 (10.15)

9. Secondary Outcome: Motor Changes Assessed With the Tinetti Test
Description: The Tinetti test is used between Visit 1 and Visits 2, 4, 5. The Tinetti test is a clinical test for the assessment of balance and gait. It has a gait score and a balance score using a 3-point ordinal scale of 0, 1 and 2. Gait is scored over 12 and balance is scored over 16 totalling 28. The lower the score on the Tinetti test, the higher the risk of falling. Tinetti test score equal or less than 18 shows high risk of fall, 19-23 scores show moderate risk of fall, and score equal or higher than 24 shows low risk of fall. Thus, min value is 0, max value is 28, higher scores mean a better outcome.
Time Frame: Day 14 (Visit 2), Day 44±2 (Visit 4), Day 75+2 (Visit 5) compared with the baseline level (Visit 1, Day 1 of treatment)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Main (Mexidol) | Control (Placebo)
Number analyzed (Participants) | 159 | 158
score on a scale
  Tinetti test, Visit 2 | 34.26 (4.92) | 34.00 (4.75)
  Difference at Visit 2 in comparison with Visit 1 | 1.62 (2.47) | 0.71 (2.84)
  Tinetti test, Visit 4 | 35.06 (4.57) | 34.39 (4.47)
  Difference at Visit 4 in comparison with Visit 1 | 2.44 (3.20) | 1.18 (3.51)
  Tinetti test, Visit 5 | 35.97 (4.26) | 34.75 (4.42)
  Difference at Visit 5 in comparison with Visit 1 | 3.36 (3.39) | 1.55 (4.05)

10. Secondary Outcome: Change in Global Illness Severity Assessed With the Clinical Global Impressions Scale at Visit 5 Compared to Baseline Measure
Description: The Clinical Global Impressions Scale is a standardized assessment tool used to rate the severity of illness, change over time, and efficacy of medication.
  The interpretation of scores is as follows:
  00 - Not assessed
  01 - Vast improvement. Side effects - None. 03 - Vast improvement. Side effects - Significantly interfere with patient's therapeutic patient's functioning 04 - Vast improvement. Side effects - outweights therapeutic effect 05 - Decided improvement. Side effects - none 09 - Slight improvement. Side effects - none 10 - Slight improvement. Side effects - do not significantly interfere with patient's functioning 13 - Slight improvement. Side effects - none
Time Frame: Day 75+2 (Visit 5)
Population: The analysis was performed for the PP-population (312 participants).
Measure: Count of Participants; unit: Participants
Arm/Group | Main (Mexidol) | Control (Placebo)
Number analyzed (Participants) | 157 | 155
Participants
  01 | 45 | 7
  03 | 1 | 0
  04 | 0 | 1
  05 | 39 | 16
  09 | 54 | 56
  10 | 3 | 0
  13 | 15 | 75

ADVERSE EVENTS:
Time Frame: From Day 1 (Visit 1) to Day 75+2 (Visit 5) or Early Termination Visit
Arm/Group | Main (Mexidol) | Control (Placebo)
All-Cause Mortality (participants affected / at risk) | 0/159 | 0/159
Serious Adverse Events (participants affected / at risk) | 0/159 | 0/159
Other Adverse Events (participants affected / at risk) | 19/159 | 32/159
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Main (Mexidol) (N=159) | Control (Placebo) (N=159)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 1 (1)
Respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Itchy nose (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Itchy throat (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Backache (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dysgeusia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 2 (2)
Leukocyturia (Renal and urinary disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Viral pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
High blood pressure (Cardiac disorders) | 0 (0) | 2 (2)
High levels of alanine aminotransferase (Investigations) | 0 (0) | 3 (3)
High levels of aspartate aminotransferase (Investigations) | 0 (0) | 2 (2)
High levels of blood creatinine (Investigations) | 0 (0) | 1 (1)
High levels of blood urea (Investigations) | 0 (0) | 1 (1)
Limb pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Balance disorder (Nervous system disorders) | 0 (0) | 1 (1)
Hematuria (Renal and urinary disorders) | 0 (0) | 2 (2)
Hyperoxaluria (Renal and urinary disorders) | 0 (0) | 1 (1)
Glycosuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal pain (Renal and urinary disorders) | 0 (0) | 1 (2)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Right bundle branch block (Cardiac disorders) | 0 (0) | 1 (1)
Heart palpitation (Cardiac disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Hyperemia (Vascular disorders) | 0 (0) | 1 (1)
Burning sensation (General disorders) | 0 (0) | 1 (2)
Panic attack (Psychiatric disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2020-04-30): https://cdn.clinicaltrials.gov/large-docs/90/NCT06834490/Prot_000.pdf
  • Statistical Analysis Plan (2020-11-06): https://cdn.clinicaltrials.gov/large-docs/90/NCT06834490/SAP_001.pdf